CLINICAL TRIAL: NCT04915768
Title: A First-in-human Phase 1 Clinical Trial to Evaluate the Safety and Immunogenicity of Stabilized CH505 TF chTrimer in Healthy, HIV-uninfected Adult Participants.
Brief Title: Evaluating the Safety and Immunogenicity of Stabilized CH505 TF chTrimer in Healthy, HIV-uninfected Adult Participants.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HVTN 300; 38705 (Registry Identifier: 38705)
Record Dates: First submitted 2021-06-01; First posted 2021-06-07 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1:Treatment (Experimental): CH505 TF chTrimer 300 mcg admixed with (5 mcg) 3M-052-AF + (500 mcg) Aluminum Hydroxide suspension, administered at months 0, 2, 4, 8 and 12.
  Interventions: Biological: CH505 TF chTrimer; Biological: 3M-05-AF; Biological: Aluminum hydroxide suspension
- Group 2: Treatment (Experimental): CH505 TF chTrimer 300 mcg admixed with (3 mcg) 3M-052-AF administered at months 0, 2, 4, 8 and 12.
  Interventions: Biological: CH505 TF chTrimer; Biological: 3M-05-AF
- Group 3: Treatment (Experimental): CH505 cTrimer, 300 mcg admixed with (3 mcg) 3M-052-AF + (500 mcg) Aluminum Hydroxide Ssuspension (Alum) administered at months 0, 2, 4, 8 and 12.
  Interventions: Biological: CH505 TF chTrimer; Biological: 3M-05-AF; Biological: Aluminum hydroxide suspension
- Group 4: Treatment (Experimental): CH505 chTrimer 300 mcg admixed with (5 mcg) 3M-052-AF administered at months 0, 2, 4, 8 and 12.
  Interventions: Biological: CH505 TF chTrimer; Biological: 3M-05-AF

INTERVENTIONS:
Biological: CH505 TF chTrimer — Combined with adjuvants 3M-052-AF and Alum. Combination administered as two 0.5 mL doses via intramuscular injection into deltoid muscle.
Biological: 3M-05-AF — Combined with CH505 TF chTrimer and Alum adjuvant. Combination administered as two 0.5 mL doses via intramuscular injection into deltoid muscle.
Biological: Aluminum hydroxide suspension — Combined with CH505 TF chTrimer and 3M-052-AF adjuvant. Combination administered as two 0.5 mL doses via intramuscular injection into deltoid muscle
  Arms: Group 1:Treatment; Group 3: Treatment

SUMMARY:
This is an open-label Phase 1 study to examine the safety and immunogenicity of the CH505 TF chTrimer vaccine with 3M-052-AF +/- Alum adjuvant in healthy adults. The primary hypothesis is that the CH505 TF chTrimer will expand CH103-like B-cell precursors.

HVTN 300 Part A examines the safety and immunogenicity of the CH505TF chTrimer with 5 mcg 3M-052-AF + 500 mcg Alum.

HVTN 300 Part B is being added to this protocol with a goal of assessing the optimal dosing and combination of 3M-052-AF and Alum adjuvant, that can potentially lead to improved neutralizing antibody activity and decreased reactogenicity, compared to Part A. Three groups have been added to Part B (Group 2: 3 mcg 3M-052-AF without Alum, Group 3: 3 mcg 3M-052 with Alum, and Group 4: 5 mcg 3M-052-AF without Alum).

DETAILED DESCRIPTION:
The primary hypothesis is that the CH505 TF chTrimer vaccine will expand B cell precursor lineages capable of ultimately producing autologous and heterologous Tier 2 broadly neutralizing antibodies (bnAbs). Participants will receive CH505 TF chTrimer plus via two intramuscular injections administered five times throughout the study. Participants will be evaluated for safety and immune responses through blood collection at specified timepoints throughout the study. Each participant will have up to 18 months of scheduled clinic visits and will have a follow-up safety assessment 12 months after their final vaccination. 3M-052-AF (at either a 3 mcg dose or a 5 mcg dose), with or without Alum, via two intramuscular injections administered five times throughout the study. Participants will be evaluated for safety and immune responses through blood collection at specified timepoints throughout the study. Each participant will have up to 18 months of scheduled clinic visits and will have a follow-up safety assessment 12 months after their final vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to complete the informed consent process, including an Assessment of Understanding: volunteer demonstrates understanding of this study; completes a questionnaire prior to first vaccination with verbal demonstration of understanding of all questionnaire items answered incorrectly.
* 18-55 years old, inclusive, on day of enrollment.
* Available for clinic follow-up through the last clinic visit, willing to undergo lymph node fine needle aspiration and leukapheresis, and willing to be contacted 12 months after the last vaccine administration.
* Agrees not to enroll in another study of an investigational agent during participation in the trial.
* In good general health according to the clinical judgement of the site investigator.
* Physical examination and laboratory results without clinically significant findings that would interfere with assessment of safety or reactogenicity in the clinical judgement of the site investigator.
* Assessed as low risk for HIV acquisition per low risk guidelines (see protocol for more information), agrees to discuss HIV infection risks, agrees to risk reduction counseling, and agrees to avoid behavior associated with high risk of HIV exposure through the final study visit. Low risk may include persons stably taking PrEP (pre- exposure prophylaxis) as prescribed for 6 months or longer.
* Hemoglobin >12.5 mg/dL to 18 mg/dL
* White blood cell (WBC) count > 3,500/mm³
* Platelets ≥125,000 /mm³
* Alanine aminotransferase (ALT) < 2.5 x ULN based on the institutional normal range
* Serum creatinine ≤1.1 x ULN based on the institutional normal range
* Blood pressure in the range of 90 to < 160 mmHg systolic and 50 to < 100 mmHg diastolic.
* Negative results for HIV infection by an FDA-approved enzyme immunoassay (EIA) or chemiluminescent microparticle immunoassay (CMIA).
* Negative for anti-Hepatitis C antibodies (anti-HCV) or negative HCV nucleic acid test (NAT) if anti-HCV antibodies are detected.
* Negative for Hepatitis B surface antigen.
* For a volunteer capable of becoming pregnant:

  * Volunteers who were assigned female sex at birth and are of reproductive potential must agree to use effective means of birth control from at least 21 days prior to enrollment through 8 weeks after their fifth vaccination timepoint (see Appendix E).
  * Has negative β-HCG (human chorionic gonadotropin) pregnancy test (urine or serum) on day of enrollment.

Exclusion Criteria:

* Volunteer who is breast-feeding or pregnant.
* Previous or current recipient of an investigational HIV vaccine (previous placebo recipients are not excluded).
* Systemic glucocorticoid use equal to or greater than prednisone10 mg/day within 3 months prior to enrollment, or other systemic medication use likely to impair immune response to vaccine in the opinion of the site investigator.
* Blood products or immunoglobulin within 16 weeks prior to enrollment; receipt of immunoglobulin within 16 weeks prior to enrollment requires PSRT approval.
* Receipt of any live attenuated vaccine within 4 weeks prior to enrollment.
* Receipt of any vaccines that are not live attenuated within 14 days prior to enrollment; replication incompetent vaccines such as the Jynneos vaccine for the prevention of monkeypox disease are not considered to be live vaccines.
* ACAM2000 vaccine for Monkeypox received within 30 days prior to enrollment or receipt of study product, or if ACAM2000 received greater than 30 days prior to enrollment or receipt of study product, vaccination scab still present; or planned administration within 30 days after enrollment or receipt of study product.
* Initiation of antigen-based immunotherapy for allergies within the previous year (stable immunotherapy is not exclusionary); inclusion of participants who initiated immunotherapy within the previous year requires PSRT approval.
* Receipt of investigational research agents with a half-life of 7 or fewer days within 4 weeks prior to enrollment. If a potential participant has received investigational agents with a half-life greater than 7 days (or unknown half- life) within the past year, PSRT approval is required for enrollment.
* Serious reactions to vaccines that preclude receipt of study injections as determined by the principal investigator or designee.
* Hereditary angioedema, acquired angioedema, or idiopathic forms of angioedema.
* Idiopathic urticaria within the past year.
* Bleeding disorder diagnosed by a doctor (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions).
* Seizure disorder; febrile seizures as a child or seizures secondary to alcohol withdrawal more than 5 years ago are not exclusionary.
* Asplenia or functional asplenia.
* Active duty and reserve US military personnel.
* Any other chronic or clinically significant condition that in the clinical judgement of the investigator would jeopardize the safety or rights of the study participant, including, but not limited to: clinically significant forms of drug or alcohol abuse, serious psychiatric disorders, or cancer that, in the clinical judgement of the site investigator, has a potential for recurrence (excluding basal cell carcinoma).
* Asthma is excluded if the participant has ANY of the following:

  * Required either oral or parenteral corticosteroids for an exacerbation two or more times within the past year; OR
  * Needed emergency care, urgent care, hospitalization, or intubation for an acute asthma exacerbation within the past year (eg, would NOT exclude individuals with asthma who meet all other criteria but sought urgent/emergent care solely for asthma medication refills or co-existing conditions unrelated to asthma); OR
  * Uses a short-acting rescue inhaler more than 2 days/week for acute asthma symptoms (ie, not for preventive treatment prior to athletic activity); OR
  * Uses medium-to-high-dose inhaled corticosteroids (greater than 250 mcg fluticasone or therapeutic equivalent per day), whether in single-therapy or dual-therapy inhalers (ie, with a long-acting beta agonist [LABA]);
  * Uses more than one medication for maintenance therapy daily. Inclusion of anyone on a stable dose of more than one medication for maintenance therapy daily for greater than two years requires PSRT approval.
* A participant with a history of an immune-mediated disease, either active or remote. Specific examples are listed in Appendix F (AESI index). Not exclusionary:

  * remote history of Bell's palsy (>2 years ago) not associated with other neurologic symptoms,
  * mild psoriasis that does not require ongoing systemic treatment
* History of allergy to local anesthetic (Novocaine, Lidocaine).
* Investigator concern for difficulty with venous access based upon clinical history and physical examination. For example, history of IV drug abuse or substantial difficulty with previous blood draws.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2023-01-23 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Frequency of CD4 binding-site-specific IgG+ B cells | Thru week 80
  Measured by flow cytometry analysis
Frequency of v2 apex and V3 glycan- specific IgG+ B cells | Thru week 80
  Measured by flow cytometry analysis
Frequency of CH505TF-specific IgG+ B cells | Thru week 80
  Measured by flow cytometry analysis
Response rate of serum antibody neutralization of vaccine-matched tier 2 HIV-1 strains | Thru week 80
  Measured by TZM-b1 assay
Magnitude of serum antibody neutralization of vaccine-matched tier 2 HIV-1 strains | Thru week 80
  Measured by TZM-b1 assay
Number of participants showing local vaccination reactogenicity signs and symptoms | 7 days following each vaccination
  Assessed by clinic staff. For a given sign or symptom, each subject's reactogenicity will be counted once under the maximum severity for each injection/ vaccination.
Number of participants showing systemic vaccination reactogenicity signs and symptoms | 7 days following each vaccination
  Assessed by clinic staff. For a given sign or symptom, each subject's reactogenicity will be counted once under the maximum severity for each injection/ vaccination.
Number of unsolicited adverse events (AEs) | 30 days following each vaccination
  Adverse events (AEs) will be graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1 (exceptions apply) for each injection/ vaccination.
Number of serious adverse events (SAEs) | Thru week 104
  Description: Adverse events (AEs) will be graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1 (exceptions apply).
Number of medically attended adverse events (MAAEs) | Thru week 104
  Description: Adverse events (AEs) will be graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1 (exceptions apply).
Number of adverse events of special interest (AESIs) | Thru week 104
  Adverse events (AEs) will be graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1 (exceptions apply).
Number of AEs leading to early participant withdrawal or permanent discontinuation | Thru week 104
  Adverse events (AEs) will be graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1 (exceptions apply).

SECONDARY OUTCOMES:
Response rate of serum IgG binding antibodies | Thru week 80
  Assessed by binding Ab multiplex assay (BAMA)
Magnitude of serum IgG binding antibodies | Thru week 80
  Assessed by binding Ab multiplex assay (BAMA)
Response rate of serum antibody neutralization of heterologous HIV-1 strains | Thru week 80
  Measured by TZM-b1 assay
Magnitude of serum antibody neutralization of heterologous HIV-1 strains | Thru week 80
  Measured by HZM-b1 assay

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth H Mayer, M.D., Study Chair — Beth Israel Deaconess Medical Center; Lindsey R Baden, M.D., Study Chair — Brigham and Women's Hospital
Locations (3):
- United States (3):
  - The Hope Clinic of the Emory Vaccine Center CRS, Decatur, Georgia
  - Brigham and Women's CRS, Boston, Massachusetts
  - Vanderbilt Vaccine (VV) CRS, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No